CLINICAL TRIAL: NCT01173809
Title: Effect of Amiodarone on the Procedure Outcome in Long-standing Persistent Atrial Fibrillation Undergoing Pulmonary Vein Antral Isolation
Acronym: SPECULATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Collaborators: University of Kansas (Other); California Pacific Medical Center (Other); Stanford University (Other); Case Western Reserve University (Other); Southlake Regional Health Centre (Other); Catholic University, Italy (Other)
Responsible Party: Principal Investigator, Andrea Natale, Medical director, Texas Cardiac Arrhythmia Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCAI-SPECULATE
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Atrial Fibrillation
Keywords: AF; Catheter Ablation; Recurrence of AF; Amiodarone
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Patient will continue taking Amiodarone before, during and after catheter ablation (8 weeks post-ablation).
  Interventions: Drug: Amiodarone
- Study (Active Comparator): Amiodarone therapy will be stopped at least 5-months before ablation procedure and ablation will be performed off Amiodarone. Patients will not take Amiodarone during the blanking period (8 weeks post-ablation).
  Interventions: Drug: Amiodarone

INTERVENTIONS:
Drug: Amiodarone — Patient will continue taking Amiodarone before, during and after ablation (8 weeks post-ablation).
  Arms: Control
Drug: Amiodarone — Amiodarone therapy will be stopped at least 5-months before ablation procedure and ablation will be performed off Amiodarone. Patients will not take Amiodarone during the blanking period (8 weeks post-ablation).
  Arms: Study

SUMMARY:
This prospective randomized study aims to investigate the effect of continuous versus interrupted use of Amiodarone on the procedure outcome in long-standing persistent (LSP) atrial fibrillation patients undergoing pulmonary vein antral isolation (PVAI).

DETAILED DESCRIPTION:
Background: Atrial Fibrillation (AF) is the most prevalent sustained clinical arrhythmia encountered in clinical practice. Its prevalence is 0.4-1% in the general population and greater than 8% in individuals >80 years of age. An estimated 2.5million individual in North America and 4.5 million in Europe are affected by AF (1). There are two fundamental principles in the management of AF; 1) anticoagulation to reduce the risk of thromboembolism, 2) ablation therapy or drugs or both to control the arrhythmia (2).

Amiodarone, a potent antiarrhythmic drug, is recommended for both atrial and ventricular arrhythmia. It has a combination of Beta-blockade, calcium-, sodium- and potassium-channel blockade effect. Most importantly, the potassium-channel blockade slows repolarization, causing an increase in the action-potential duration and in the refractoriness of the cardiac musculature (3). As the myocardium remains unresponsive, the premature depolarizations which were previously causing AF are prevented from propagation.

During the ablation procedure, mapping electrograms using circular mapping catheter and provocative maneuvers such as administration of isoproterenol in incremental doses are commonly used to aid in identification of pulmonary vein (PV) and non-PV triggers. In addition, areas with complex fractionated atrial electrograms (CFAE) are identified and eliminated by ablation. In patients with LSP, inclusion of PV and non-PV triggers as ablation targets, improves the procedure outcome.

As Amiodarone increases the refractoriness of the myocardium, it is possible that under the effect of Amiodarone some of the focal triggers could be masked or remain unidentified during mapping or isoproterenol-provocation. These unrecognized triggers could cause recurrence of AF during the post-ablation period. In other words, discontinuation of Amiodarone at least 5-months before ablation could result in unmasking of all the focal triggers that would have otherwise stayed unrecognized and eliminating those triggers would significantly improve the success rate of the procedure.

Our study aims to investigate the role of Amiodarone in influencing the procedure outcome in LSP-AF patients undergoing catheter ablation.

Hypothesis: Withdrawal of Amiodarone 4 months before procedure results in unmasking of additional focal triggers, ablation of which leads to an improved procedure outcome in LSP_AF patients.

Inclusion Criteria:

1. History of LSP AF
2. Age > 18 years
3. Willing and ability to understand and sign an informed consent
4. Patients on chronic Amiodarone therapy (≥ 3 months)

Exclusion Criteria:

1. Unstable angina
2. Concomitant treatment with other class I or III antiarrhythmic drugs
3. Myocardial infarction within past 3 months)
4. Presence of any disease that is likely to shorten life expectancy to < 1 year
5. Symptomatic heart failure, NYHA III or IV
6. Contraindications for Amiodarone
7. Chronic liver diseases
8. Pregnant or breast-feeding mothers

Primary Outcome Measure:

Recurrence of AF, atrial flutter or atrial tachycardia

Secondary Outcome Measures:

Difference in the occurrence of relapse between the control and the study groups

Study design:

This is a multi-center, prospective study in which consecutively enrolled patients treated with Amiodarone for long standing persistent AF will be randomized to either the study or the control group.

Study group: Amiodarone therapy will be stopped at least 4-months before ablation procedure and ablation will be performed off Amiodarone. Patients will not take Amiodarone during the blanking period (8 weeks post-ablation).

Control group: Patient will continue taking Amiodarone before, during and after ablation (8 weeks post-ablation).

After the blanking period, everybody would be off Amiodarone unless they have recurrence. Anti-arrhythmic drugs other than Amiodarone would be tried if patient develops recurrence and repeat ablation would be considered.

Follow-Up:

Patients will be followed up for 3 years post-ablation. An ECG and telemetry transmission monitor report will be obtained in all patients at each follow-up examination.

Patients will be supplied with an Event Recorder for trans-telephonic rhythm transmission (telemetry) for 5 months after ablation, and will be asked to transmit their rhythm data every time they had symptoms compatible with arrhythmias; and at least once a week, even if they were asymptomatic. Holter monitoring will be performed at 6-month post-ablation. The arrhythmic episodes will be documented based on ECG, Holter data, Event Recorder data and/or implanted device data (when available).

In case of recurrence, if patients undergo repeat ablations, all procedures will happen off amiodarone. After redo, patients will be followed up for 1 year for recurrence in the same way as described above.

ELIGIBILITY:
Inclusion Criteria:

1. History of LSP AF
2. Age > 18 years
3. Willing and ability to understand and sign an informed consent
4. Patients on chronic Amiodarone therapy (≥ 3 months)

Exclusion Criteria:

1. Unstable angina
2. Concomitant treatment with other class I or III antiarrhythmic drugs
3. Myocardial infarction within past 3 months)
4. Presence of any disease that is likely to shorten life expectancy to < 1 year
5. Symptomatic heart failure, NYHA III or IV
6. Contraindications for Amiodarone
7. Chronic liver diseases
8. Pregnant or breast-feeding mothers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2010-10; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Recurrence of atrial arrhythmia | 1 year
  Recurrence of AF, atrial flutter or atrial tachycardia

SECONDARY OUTCOMES:
Relapse of AF | 1 yeay
  Difference in the occurrence of relapse between the control and the study groups

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, MD, Principal Investigator — TCAI, St.David's Medical Center; Luigi Di Biase, Md, PhD, Principal Investigator — Texas Cardiac Arrhythmia Research Foundation
Locations (1):
- St.David's Medical Center, Austin, Texas, United States

REFERENCES:
- [Derived] Mohanty S, Di Biase L, Mohanty P, Trivedi C, Santangeli P, Bai R, Burkhardt JD, Gallinghouse JG, Horton R, Sanchez JE, Hranitzky PM, Zagrodzky J, Al-Ahmad A, Pelargonio G, Lakkireddy D, Reddy M, Forleo G, Rossillo A, Themistoclakis S, Hongo R, Beheiry S, Casella M, Dello Russo A, Tondo C, Natale A. Effect of periprocedural amiodarone on procedure outcome in patients with longstanding persistent atrial fibrillation undergoing extended pulmonary vein antrum isolation: results from a randomized study (SPECULATE). Heart Rhythm. 2015 Mar;12(3):477-483. doi: 10.1016/j.hrthm.2014.11.016. Epub 2014 Nov 18. PMID 25460855